CLINICAL TRIAL: NCT07349550
Title: AtWork: The Relation Between Cognitive Functioning, Common Mental Disorders and Work Functioning
Acronym: AtWork
Status: Recruiting | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Diakonhjemmet Hospital (Other); The Research Council of Norway (Other)
Responsible Party: Sponsor
Other Study IDs: AtWork
Record Dates: First submitted 2025-06-17; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Depression - Major Depressive Disorder; Anxiety
Keywords: Metacognitive therapy; Work focus; Depression; Anxiety; Sick leave
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients referred with depression and/or anxiety and at risk of sick leave: Patients referred with depression and/or anxiety and at risk of sick leave

SUMMARY:
Depression and anxiety affects levels of function across different levels like work, increasing levels of sick leave and as well as cognitive functioning. In the current study patients at risk of sick leave with depression and anxiety receive metacognitive therapy and work focus in an ordinary outpatient clinic. Impaired cognitive functioning may also be of importance in the return to work process and degree of sick leave. It is important to get a better understanding of how cognitive functioning is related to sick leave and if it predicts return to work, and if cognitive functioning is changed due to psychological treatment.

DETAILED DESCRIPTION:
The study is a naturalistic study exploring cognitive functioning of patients with common mental disorders (CMD) treated with metacognitive therapy and work focused interventions, and changes over time.

Sick leave is common for patients with CMD, also after having completed treatment for CMD. Why patients remain on sick leave after having completed treatment is underexplored. Potential reasons may be that work and sick leave is not addressed during therapy, there could be issues related to the work place, also there may be characteristics related to the patients functioning that is underexplored. In the latter context, little knowledge regarding the relations between cognitive functioning, symptoms of CMD and work functioning. Previous studies have investigated neuropsychological functions in relation to work related stress and stress-related exhaustion, and found worse performance on cognitive tasks compared to healthy controls. Although stress-related exhaustion can be considered a phenomenon related to CMD, there are no studies the investigators are aware of that investigate neuropsychological predictors specifically related to CMD and work functioning. A review from 2022 specifically aimed to identify neuropsychological predictors of vocational rehabilitation outcomes in individuals with MDD specifically, and found no studies. This clearly demonstrates a knowledge gap that this project would fill. E.g., lower cognitive functioning after successful treatment of CMD is related to increased risk of additional sick leave. With this in mind, increasing our knowledge of these variables can help clinicians identify patients at risk for additional sick leave, even after successful treatment. A previous study at the same clinic has identified three subgroups in a sample of patients with CMD at risk of sick leave. The first group was never on sick leave. The second group returned to work after sick leave during or shortly after treatment. In the third group half of the patients remained on sick leave or disability. To better understand characteristics of such subgroups it is relevant to explore standard clinical information given in the patient's journal. This project is mainly, but not exclusively a PhD-project. The time schedule for the project will go beyond the time for the PhD, especially long-time follow-up.

The main aims of the project are the following:

To explore how descriptive variables, CMD symptoms, and cognitive functioning are associated with work functioning (sick leave or risk for sick leave) before treatment. And what is the interplay between symptoms, cognitive profiles and sick leave.

To explore whether cognitive functioning can predict outcomes of both symptoms of CMD and degree of sick leave, and if cognitive functioning changes through MCT and work focused interventions.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of depression and/or anxiety,
* at risk of sick leave

Exclusion Criteria:

* personality disorders cluster A or B,
* ongoing substance abuse,
* symptoms of psychosis,
* acute suicidality,
* serious somatic disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred with depression and/or anxiety disorders at risk of sick leave.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2029-08-01 (Estimated); Study Completion 2032-08-01 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Measured at pre-treatment and at therapy completion, an average of 10 weekly sessions, and at 6, 12 months follow-up
  Measure of depressive symptoms (PHQ-9) range 0-27 higher scores indicate higher degree of depressive symptoms
Generalized Anxiety Disorder (GAD-7) | Measured at pre-treatment and at therapy completion, an average of 10 weekly sessions, and at 6, 12 months follow-up
  Anxiety symptoms (GAD-7) range 0-21 higher scores indicating higher degree of anxiety symptoms
Changes in sick leave | Measured at pre-treatment and at therapy completion, an average of 10 weekly sessions, and at 6, 12 months follow-up
  Sick leave is collected from national register data measured in number of days of sick leave.

CONTACTS AND LOCATIONS:
Locations (1):
- Diakonhjemmet hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Due to ethical considerations as this is a clinical study that includes patients with depression and/or anxiety at risk of sick leave, information will not be shared